CLINICAL TRIAL: NCT05537233
Title: Efficacy and Safety of Once Weekly Semaglutide in Adults With Obesity and Inadequately Controlled Type 1 Diabetes Using Hybrid Closed-Loop System.
Brief Title: ADJUnct Semaglutide Treatment in Type 1 Diabetes
Acronym: ADJUST-T1D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viral N. Shah (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Viral N. Shah, Professor of Medicine, Division of Endocrinology & Metabolism, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22388
Record Dates: First submitted 2022-08-23; First posted 2022-09-13 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes; Obesity
Keywords: Type 1 diabetes; Obesity; HbA1c; Time-in-range; Weight loss; Cardiovascular risk
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Obesity; Weight Loss | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Participants in this group will receive semaglutide once weekly injection in addition to their standard closed-loop therapy
  Interventions: Drug: Semaglutide
- Control (Placebo Comparator): Participants in this group will receive placebo once weekly injection in addition to their standard closed-loop therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Semaglutide up to 1 mg per week in addition to standard closed-loop therapy
  Arms: Semaglutide
Drug: Placebo — Injection placebo up to 1 mg per week in addition to standard closed-loop therapy
  Arms: Control

SUMMARY:
The purpose of this study is to assess the use of once weekly semaglutide injection in inadequately controlled obese adults with type 1 diabetes (T1D) using FDA-approved hybrid closed-loop therapies.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients given written informed consent will undergo a 2-week screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized in a double-blind manner using computer generated randomization scheme to receive either semaglutide or placebo (1:1 ratio) for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

For an eligible subject, all inclusion criteria must be answered "yes"

1. Age ≥18 and ≤ 65 years
2. Patients with clinical diagnosis of T1D diagnosed for at least 12 months
3. Patient is on FDA- approved hybrid closed-loop system for ≥ 3 months
4. Willing to use once weekly semaglutide
5. Willing to share devices (HCL system) data uploads
6. HbA1c >7.0% and <10.0%
7. Body mass index ≥30 kg/m2
8. Has current glucagon product to treat severe hypoglycemia
9. Has current ketone meters to check ketones
10. Ability to provide informed consent before any trial-related activities

Exclusion Criteria:

1. Age <18 years and >65 years
2. HbA1c ≤7.0 % or ≥ 10.0% at screening
3. Less than 12 months of insulin treatment
4. Use of unapproved insulin for HCL system. E.g. use of Fiasp in the Tandem Control-IQ system
5. Not willing to share the devices (HCL system) data uploads
6. Non compatible devices (e.g. pump, CGM or smart phones) for data transfer
7. Current use of multiple daily injection or inhaled insulin (Afrezza)
8. Patients with T1D using any glucose lowering medications other than insulin at the time of screening
9. Pregnancy, breast feeding, and positive pregnancy test during screening
10. Women of childbearing age wanting to become pregnant
11. Unwilling to use acceptable contraceptive methods (for both men and women) during the trial period
12. Current use (≥ 2 weeks of continuous use) of any steroidal medication, or anticipated long-term steroidal treatment (>4 weeks continuously), during the study period
13. Use of GLP-1RA or weight loss medications in the past 3 month
14. Clinical diagnosis/history of gastroparesis or gastric motility disorders
15. Serum triglycerides >500 mg/dL
16. Planning for bariatric surgery during the study period
17. eGFR below 45 ml/min/1.73 m^2 using CKD-EPI formula
18. History of severe hypoglycemia in the previous 3 months
19. History of diabetic ketoacidosis requiring hospitalization in the past 3 months
20. History of allergy to any form of insulin, GLP-1RA or its excipients
21. History of any form of pancreatitis
22. History of stroke, myocardial infarction in the past 3 months
23. History of congestive heart failure class III or IV
24. History of acute or chronic liver disease
25. History of malignancy requiring chemotherapy, surgery or radiation in previous 5 years
26. Personal or family history of multiple endocrine neoplasia type 2 (MEN-2) or familial thyroid carcinoma or non-familial medullary thyroid carcinoma
27. Have a pacemaker, metal implants, or aneurysm clips or weigh >330 lbs (exclusion only if doing MRI)
28. Use of investigational drugs within 5 half-lives prior to screening
29. Participation to other intervention trials during the study period
30. Any comorbidities or medical conditions such as severe psychiatric disorder that make a person unfit for the study at the discretion of the investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Viral N Shah, MD, Principal Investigator — Indiana University
Locations (4):
- United States (4):
  - Barbara Davis Center for Diabetes, Aurora, Colorado
  - Iowa Diabetes Research Center, West Des Moines, Iowa
  - Henry Ford Hospital, Detroit, Michigan
  - Harold Schnitzer Diabetes Health Center, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No
IPD may be available once the study is completed and all results are published.

REFERENCES:
- [Derived] Shah VN, Akturk HK, Kruger D, Ahmann A, Bhargava A, Bakoyannis G, Pyle L, Snell-Bergeon JK. Semaglutide in Adults with Type 1 Diabetes and Obesity. NEJM Evid. 2025 Aug;4(8):EVIDoa2500173. doi: 10.1056/EVIDoa2500173. Epub 2025 Jun 23. PMID 40550013

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Semaglutide | Control
Started | 36 | 36
Completed | 34 | 33
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide | Control | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (11.6) | 38.9 (13.1) | 40 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 14 | 16 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 35 | 32 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 33 | 30 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
body mass index [Mean (Standard Deviation); unit: kg/m2] | 34.7 (3.9) | 36.0 (5.2) | 35 (4.5)
HbA1c [Mean (Standard Deviation); unit: %] | 7.8 (0.6) | 7.7 (0.6) | 7.8 (0.6)
Diabetes Duration [Mean (Standard Deviation); unit: years] | 23.4 (11.2) | 21.9 (11.6) | 23 (11)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Adults With T1D Achieving Composite Outcome (CGM-measured Time in Range (TIR)>70% With Time Below Range (TBR) of <4% and Reduction in Body Weight by 5%) at 26 Weeks in the Semaglutide Group Compared to Placebo Group
Description: Primary outcome will be analyzed per statistical analysis plan using intention to treat basis.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Control
Number analyzed (Participants) | 36 | 36
Participants | 13 | 0

2. Secondary Outcome: Change in HbA1c
Description: HbA1c will be measured at a central laboratory and change in Hba1c from baseline to 26 weeks will be compared by randomization group using intention to treat (ITT) analysis.
Time Frame: 26 weeks
Measure: Least Squares Mean (Standard Error); unit: percentage HbA1c
Arm/Group | Semaglutide | Control
Number analyzed (Participants) | 36 | 36
percentage HbA1c | -0.7 (0.1) | -0.4 (0.1)

3. Secondary Outcome: Change in Mean Glucose
Description: Mean glucose (mg/dL) will be obtained by CGM and change in mean CGM glucose from baseline to 26 weeks will be compared by randomization group using intention to treat (ITT) analysis.
Time Frame: 26 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Semaglutide | Control
Number analyzed (Participants) | 36 | 36
mg/dL | -15.7 (2.6) | -3.6 (2.8)

4. Secondary Outcome: Percent Time Spent in CGM-measured Glucose Range of 70-140 mg/dL (Time in Tight Target Range; TTIR)
Description: Percent of time spent in tight glucose range (70-140 mg/dL) will be obtained by CGM and change in percent time in range from baseline to 26 weeks will be compared by randomization group using intention to treat (ITT) analysis.
Time Frame: 26 weeks
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Arm/Group | Semaglutide | Control
Number analyzed (Participants) | 36 | 36
percentage of time | 9.8 (1.7) | 2.9 (1.8)

5. Secondary Outcome: Percent Time Spent in CGM-measured Glucose >180 mg/dL
Description: Percent of time spent in glucose range >180 mg/dL will be obtained by CGM and change in mean CGM glucose from baseline to 26 weeks will be compared by randomization group using intention to treat (ITT) analysis.
Time Frame: 26 weeks
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Semaglutide | Control
Number analyzed (Participants) | 36 | 36
percentage | -11.1 (1.8) | -2.7 (1.9)

6. Secondary Outcome: Percent Time Spent in CGM-measured Glucose >250mg/dL
Description: Percent of time spent in glucose range >250 mg/dL will be obtained by CGM and change in mean CGM glucose from baseline to 26 weeks will be compared by randomization group using intention to treat (ITT) analysis.
Time Frame: 26 weeks
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Semaglutide | Control
Number analyzed (Participants) | 36 | 36
percentage | -5.1 (1.1) | -0.5 (1.2)

7. Secondary Outcome: Percent Time Spent in CGM-measured Glucose <70mg/dL
Description: Percent of time spent in glucose range <70 mg/dL will be obtained by CGM and change in mean CGM glucose from baseline to 26 weeks will be compared by randomization group using intention to treat (ITT) analysis.
Time Frame: 26 weeks
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Semaglutide | Control
Number analyzed (Participants) | 36 | 36
percentage | 0.1 (0.2) | 0.4 (0.2)

8. Secondary Outcome: Change in CGM Measured Glycemic Variability (Coefficient of Variation)
Description: Glucose coefficient of variation (mg/dL) will be obtained by CGM and change in glucose CV from baseline to 26 weeks will be compared by randomization group using intention to treat (ITT) analysis.
Time Frame: 26 weeks
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Semaglutide | Control
Number analyzed (Participants) | 36 | 36
percentage | -0.3 (0.8) | 0.9 (0.9)

9. Secondary Outcome: Change in Weight
Description: The change in kg of body weight from baseline to 26 weeks will be compared by randomization group using an ITT analysis.
Time Frame: 26 weeks
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Semaglutide | Control
Number analyzed (Participants) | 36 | 36
kg | -9.2 (0.7) | -0.4 (0.6)

10. Secondary Outcome: Change in BMI (Kg/m2)
Description: Change in body mass index (BMI) calculated as kg body weight per meter squared of height from baseline to 26 weeks will be compared by randomization group using an ITT analysis.
Time Frame: 26 weeks
Measure: Least Squares Mean (Standard Error); unit: kg/m2
Arm/Group | Semaglutide | Control
Number analyzed (Participants) | 36 | 36
kg/m2 | -3.3 (0.3) | -0.2 (0.2)

11. Secondary Outcome: Severe Hypoglycemia
Description: SH events in number of patients per group
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Control
Number analyzed (Participants) | 36 | 36
Participants | 2 | 2

12. Other Pre Specified Outcome: Change in Patient Reported Quality of Life
Description: Patient reported quality of life will be measured using a validated instrument (ADDQOL) and the change in score from baseline to 26 weeks will be compared by randomization group using an ITT analysis.
Time Frame: 26 weeks
Reporting Status: Not Posted, anticipated posting 2026-07

13. Other Pre Specified Outcome: Proportion of Participants With HbA1c <7%
Description: proportion (N, %) of participants achieving HbA1c <7% between two groups over 26 weeks
Time Frame: 26 weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Proportion of Participants With HbA1c <7.5%
Description: proportion (N, %) of participants achieving HbA1c <7.5% between two groups over 26 weeks
Time Frame: 26 weeks
Reporting Status: Not Posted

15. Other Pre Specified Outcome: HbA1c Improvement
Description: HbA1c improvement from baseline to 26 weeks between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: HbA1c Improvement of >0.4% From Baseline
Description: proportion of participants with HbA1c improvement of >0.4% from baseline between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Proportion of Participants Achieving TIR >70%
Description: Proportion of participants achieving TIR >70% between two groups over 26 weeks
Time Frame: 26 weeks
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Proportion of Participants Achieving TITR >50%
Description: Proportion of participants achieving TITR (time in 70-140 mg/dL) >50% between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Proportion of Participants Achieving TIR >80%
Description: Proportion of participants achieving TIR >80% between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Proportion of Participants Achieving TITR >60%
Description: Proportion of participants achieving TITR (time in 70-140 mg/dL) >60% between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Number of TBR<70 Events
Description: Numbers of events of CGM glucose <70 mg/dL lasting for at least 15 minutes between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Number of TBR <54 Events
Description: Numbers of events of CGM glucose <54mg/dL lasting for at least 15 minutes between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Change in Total Daily Dose of Insulin (TDD, Units Per Day and U/Kg/Day)
Description: Change in TDD between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Proportion Achieving Weight Loss ≥5%
Description: Proportion of participants achieving weight loss ≥5% from baseline between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Proportion Achieving Weight Loss ≥10%
Description: Proportion of participants achieving weight loss ≥10% from baseline between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Proportion of Achieving BMI <30 kg/m2
Description: Proportion of participants achieving BMI <30 kg/m2 between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Proportion of Achieving BMI <25 kg/m2
Description: Proportion of participants achieving BMI <25 kg/m2 between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Change in Systolic Blood Pressure (SBP)
Description: change in SBP (mmHg) between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Change in Diastolic Blood Pressure (DBP)
Description: change in DBP (mmHg) between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Change in Pulse Pressure
Description: change in pulse pressure between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Change in Triglyceride/HDL Ratio
Description: Change in triglyceride/HDL ratio between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Change in Brach D
Description: Change in brachial arterial distensibility between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Change in Carotid Intima Media Thickness (cIMT)
Description: Change in carotid intima media thickness (cIMT) between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Change in Femoral to Carotid Pulse Wave Velocity (m/s)
Description: Change in femoral to carotid pulse wave velocity (m/s) between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Change in Urine Albumin to Creatinine Ratio (ACR)
Description: Change in ACR between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Quality of Life (Diabetes Dependent QOL)
Description: Change in QOL between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Change in CGM Metrics by Daytime vs Nighttime
Description: Change in CGM metrics (TIR, TITR, mean glucose, TBR, TAR >180, SD, CV) by daytime (6 AM to <11 PM) and nighttime (11 PM to <6 AM) between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

38. Other Pre Specified Outcome: AID Setting Adjustment
Description: Defined any adjustment in settings by provider or patient per person over the study period by two groups (number of adjustments (N) during trial) between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Change in Basal Insulin Per Day
Description: Change in basal insulin per day (Total basal insulin including autobasal delivery, units per day and U/kg/day) between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

40. Other Pre Specified Outcome: Change in Total Boluses Per Day
Description: Change in total boluses per day (frequency of boluses per day) between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

41. Other Pre Specified Outcome: Achievement of Primary Outcome and Key Secondary Outcomes by Types of AID Systems
Description: Proportion of participants achieving primary outcome and key secondary glycemic outcomes by types of AID systems
Time Frame: 26 weeks
Reporting Status: Not Posted

42. Other Pre Specified Outcome: Change in Carbohydrate Intake Per Day (Grams/Day)
Description: Change in Carbohydrate intake per day (grams/day) between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

43. Other Pre Specified Outcome: Change in Total Bolus Insulin Per Day
Description: Change in total bolus insulin per day (units per day and U/Kg/day) between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

44. Other Pre Specified Outcome: Change in eGFR
Description: Change in eGFR using CKD-EPI between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

45. Other Pre Specified Outcome: Change in Fib-4 Score
Description: Change in Fib-4 score between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

46. Other Pre Specified Outcome: Change in HSI (Hepatic Steatosis Index)
Description: Change in HSI (hepatic steatosis index) between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

47. Other Pre Specified Outcome: Change in MRI Measured Pulse Wave Velocity and Longitudinal Strain
Description: Change in MRI measured pulse wave velocity and longitudinal strain between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

48. Other Pre Specified Outcome: Change in LDL-C
Description: Change in LDL-C between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

49. Other Pre Specified Outcome: Change in TC
Description: Change in TC between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

50. Other Pre Specified Outcome: Change in TG
Description: Change in TG between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

51. Other Pre Specified Outcome: Change in HDL-C
Description: Change in HDL-C between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

52. Other Pre Specified Outcome: Proportion With ACR <30 at 26 Weeks
Description: Proportion of participants with ACR <30 at 26 weeks between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

53. Other Pre Specified Outcome: Proportion With Change in ACR From >30 to <30
Description: Proportion of participants with change in ACR from >30 to <30 between two groups
Time Frame: 26 weeks
Reporting Status: Not Posted

54. Other Pre Specified Outcome: Achievement of Primary Outcomes by Baseline BMI (BMI <35 vs >35)
Description: Achievement of primary outcomes by baseline BMI (BMI <35 vs >35)
Time Frame: 26 weeks
Reporting Status: Not Posted

55. Other Pre Specified Outcome: Achievement of Primary Outcomes by Baseline A1c (A1c <7.5% vs >7.5%)
Description: Achievement of primary outcomes by baseline A1c (A1c <7.5% vs >7.5%)
Time Frame: 26 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: from signing consent from till end of the study (i.e 26 weeks)
Arm/Group | Semaglutide | Control
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/36 | 0/36
Other Adverse Events (participants affected / at risk) | 26/36 | 11/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide (N=36) | Control (N=36)
Nausea & vomiting (Gastrointestinal disorders) | 1 (1) | 0 — Severe GI event leading to hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide (N=36) | Control (N=36)
Gastrointestinal events (Gastrointestinal disorders) | 19 (57) | 9 (13) — GI event: nausea, vomiting, reflux (gastrointestinal reflux disease), burping or belching, diarrhea, constipation, loss of appetite, and elevated levels of liver enzymes.
Upper respitory infectin (Infections and infestations) | 3 (4) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT05537233/Prot_SAP_001.pdf